CLINICAL TRIAL: NCT01231334
Title: A Study Comparing Aczone® Plus Differin® Versus Duac® Plus Differin® in Patients With Severe Facial Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA-ACZ1001
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone; Adapalene; Gels; Clindamycin; Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aczone® Gel 5% plus Differin® 0.3% Gel (Active Comparator): Dapsone (Aczone® Gel 5%) applied to entire face in the morning. Adapalene (Differin® 0.3% Gel)followed by Dapsone (Aczone® Gel 5%) applied to entire face in the evening. Daily treatment for 12 weeks.
  Interventions: Drug: Dapsone plus Adapalene
- Duac® Topical Gel plus Differin® 0.3% Gel (Active Comparator): Clindamycin/benzoyl peroxide (Duac® Topical Gel)applied to entire face in the morning. Adapalene (Differin® 0.3% Gel) applied to entire face in the evening. Daily treatment for 12 weeks.
  Interventions: Drug: Clindamycin/benzoyl peroxide plus Adapalene

INTERVENTIONS:
Drug: Dapsone plus Adapalene — Dapsone (Aczone® Gel 5%) applied to entire face in the morning. Adapalene (Differin® 0.3% Gel)followed by Dapsone (Aczone® Gel 5%) applied to entire face in the evening. Daily treatment for 12 weeks.
  Other Names: Aczone® Gel 5%; Differin® 0.3% Gel
  Arms: Aczone® Gel 5% plus Differin® 0.3% Gel
Drug: Clindamycin/benzoyl peroxide plus Adapalene — Clindamycin/benzoyl peroxide (Duac® Topical Gel)applied to entire face in the morning. Adapalene (Differin® 0.3% Gel) applied to entire face in the evening. Daily treatment for 12 weeks
  Other Names: Duac® Topical Gel; Differin® 0.3% Gel
  Arms: Duac® Topical Gel plus Differin® 0.3% Gel

SUMMARY:
A study comparing the topical application of Aczone® plus Differin® versus Duac® plus Differin® in patients with severe facial acne (facial acne vulgaris).

ELIGIBILITY:
Inclusion Criteria:

* Severe facial acne (acne vulgaris)

Exclusion Criteria:

* History of significant anemia or hemolysis
* History of enteritis (eg, regional enteritis, ulcerative colitis, pseudomembranous colitis, antibiotic-associated colitis)
* History of lupus, rosacea, or seborrheic dermatitis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 286 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Miramar, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aczone® Gel 5% Plus Differin® 0.3% Gel | Duac® Topical Gel Plus Differin® 0.3% Gel
Started | 145 | 141
Completed | 126 | 120
Not Completed | 19 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aczone® Gel 5% Plus Differin® 0.3% Gel | Duac® Topical Gel Plus Differin® 0.3% Gel | Total
Number analyzed (Participants) | 145 | 141 | 286
Age Continuous [Mean (Standard Deviation); unit: Years] | 27.2 (6.5) | 27.9 (7.1) | 27.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 141 | 286
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Global Acne Assessment Score (GAAS) at Week 12
Description: GAAS was conducted by the investigator. The patient's facial acne was evaluated on a 5 point scale 0=None (no evidence of acne), 1=Minimal (few lesions), 2=Mild (several to many non-inflammatory lesions; few inflammatory lesions), 3=Moderate (many lesions) to 4=Severe (Significant degree of inflammatory disease; papules/pustules present, few nodulo-cystic lesions; comedones may be present). Papules and nodules are round, solid elevations of the skin with no visible fluid. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: Per-Protocol Population consists of all randomized participants who completed the study to week 12 without any major protocol violation.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Aczone® Gel 5% Plus Differin® 0.3% Gel | Duac® Topical Gel Plus Differin® 0.3% Gel
Number analyzed (Participants) | 122 | 118
Score on a scale
  Baseline | 2.80 (0.51) | 2.84 (0.45)
  Change from baseline at Week 12 | -0.87 (0.82) | -1.27 (0.82)

2. Secondary Outcome: Percentage of Participants at Week 12 Having at Least a One Point Decrease in Overall Disease Severity
Description: The overall disease severity was evaluated by the investigator at Baseline and Week 12 using a 7-point scale to rate the overall acne severity (lesions, inflammation, facial redness and skin condition), where 0=no acne lesions and 6=most severe acne. The percentage of participants with at least a one point decrease (improvement) from baseline is calculated.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aczone® Gel 5% Plus Differin® 0.3% Gel | Duac® Topical Gel Plus Differin® 0.3% Gel
Number analyzed (Participants) | 122 | 118
Percentage of participants | 83.5 | 92.4

3. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Counts at Week 12
Description: Percent Change from baseline in inflammatory lesion counts (papules, pustules and nodules) at week 12. Papules and nodules are round, solid elevations of the skin with no visible fluid; papules are smaller (less than 5 or 10 millimeters in width and depth) and nodules are larger (greater than 5 or 10 millimeters in width and depth). Pustules are small elevations of the skin containing cloudy material. A negative number change from baseline indicates a reduction in lesion counts (improvement).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change
Arm/Group | Aczone® Gel 5% Plus Differin® 0.3% Gel | Duac® Topical Gel Plus Differin® 0.3% Gel
Number analyzed (Participants) | 122 | 118
Percent change | -70.7 [-100.0 to 38.1] | -75.9 [-100.0 to -17.4]

4. Secondary Outcome: Percent Change From Baseline in Non-inflammatory Lesion Counts at Week 12
Description: Percent Change from baseline in non-inflammatory lesion counts (open/closed comedones) at week 12. Comedones are small bumps on the skin (lesions) caused by acne and found at the opening of a skin pore. Open comedones (also known as a blackheads) have a microscopic opening to the skin surface, while closed comedones (also known as whiteheads or "pimples") lack the opening to the skin. A negative number change from baseline indicates a reduction in lesion counts (improvement).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change
Arm/Group | Aczone® Gel 5% Plus Differin® 0.3% Gel | Duac® Topical Gel Plus Differin® 0.3% Gel
Number analyzed (Participants) | 122 | 118
Percent change | -55.3 [-100.0 to 115.0] | -60.7 [-100.0 to 31.6]

5. Secondary Outcome: Percent Change From Baseline in Total Lesion Count at Week 12
Description: Percent change in total lesion counts: inflammatory (papules, pustules and nodules) and non-inflammatory (comedones) lesion counts from baseline. Papules and nodules are round, solid elevations of the skin with no visible fluid; papules are smaller (less than 5 or 10 millimeters ) and nodules are larger (greater than 5 or 10 millimeters). Pustules are small elevations of the skin containing cloudy material. Comedones are small bumps on the skin caused by acne and found at the opening of a skin pore. A negative change from baseline indicates a reduction in lesion counts (improvement).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change
Arm/Group | Aczone® Gel 5% Plus Differin® 0.3% Gel | Duac® Topical Gel Plus Differin® 0.3% Gel
Number analyzed (Participants) | 122 | 118
Percent change | -62.7 (27.0) [-98.0 to 75.6] | -65.0 (22.5) [-100.0 to 8.5]

6. Secondary Outcome: Percentage of Participants Demonstrating a ≥ 1 Category Increase in Tolerability From Baseline at Week 12
Description: The investigator rated the patient's current symptoms of erythema, dryness, peeling, and oiliness on a 5 point scale from 0 (Absent) to 4 (Severe). The investigator rated the symptoms of pruritus and burning since last visit on a 6 point scale of 0 (Absent) to 5 (Severe)-interfering with daily activities. Percentage of participants demonstrating a ≥1 category increase (improvement) in tolerability from baseline is calculated.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aczone® Gel 5% Plus Differin® 0.3% Gel | Duac® Topical Gel Plus Differin® 0.3% Gel
Number analyzed (Participants) | 122 | 118
Percentage of participants
  Dryness | 21.3 | 11.9
  Peeling | 11.5 | 9.3
  Oiliness | 6.7 | 6.0
  Erythema | 8.2 | 6.8
  Pruritus | 12.4 | 8.5
  Burning | 13.2 | 12.7

7. Primary Outcome: Percentage of Participants With at Least a One Point Decrease in the Global Acne Assessment Score (GAAS) at Week 12
Description: GAAS was conducted by the investigator at Baseline and Week 12. The patient's facial acne was evaluated on a 5 point scale 0=None (no evidence of acne), 1=Minimal (few lesions), 2=Mild (several to many non-inflammatory lesions; few inflammatory lesions), 3=Moderate (many lesions) to 4=Severe (Significant degree of inflammatory disease; papules/pustules present, few nodulo-cystic lesions; comedones may be present). Papules/nodules are round, solid elevations of the skin with no visible fluid. The percentage of participants with at least a one point decrease (improvement) in GAAS was calculated.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aczone® Gel 5% Plus Differin® 0.3% Gel | Duac® Topical Gel Plus Differin® 0.3% Gel
Number analyzed (Participants) | 122 | 118
Percentage of participants | 69.7 | 81.4

ADVERSE EVENTS:
Description: Safety population includes all participants who received study treatment.
Arm/Group | Aczone® Gel 5% Plus Differin® 0.3% Gel | Duac® Topical Gel Plus Differin® 0.3% Gel
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/135
Other Adverse Events (participants affected / at risk) | 23/136 | 15/135
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aczone® Gel 5% Plus Differin® 0.3% Gel (N=136) | Duac® Topical Gel Plus Differin® 0.3% Gel (N=135)
Nasopharyngitis (Infections and infestations) | 15 | 7
Headache (Nervous system disorders) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.